CLINICAL TRIAL: NCT00994292
Title: A Randomized, Double-Blind, Placebo Controlled Multi-Center and Parallel Group Study of the Safety, Tolerability and Efficacy of YM150 in Combination With Standard Treatment in Secondary Prevention of Ischemic Vascular Events in Subjects With Acute Coronary Syndromes
Brief Title: Study Evaluating Safety, Tolerability and Efficacy of YM150 in Subjects With Acute Coronary Syndromes
Acronym: RUBY-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 150-CL-201; 2008-005972-29 (EudraCT Number)
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-09

CONDITIONS: Acute Coronary Syndrome
Keywords: Factor Xa; Anticoagulant; YM150; Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- 1. YM150 Dose V, twice daily (Experimental)
  Interventions: Drug: YM150
- 2. YM150 Dose W, once daily (Experimental)
  Interventions: Drug: YM150
- 3. YM150 Dose X, twice daily (Experimental)
  Interventions: Drug: YM150
- 4. YM150 Dose Y, once daily (Experimental)
  Interventions: Drug: YM150
- 5. YM150 Dose Y, twice daily (Experimental)
  Interventions: Drug: YM150
- 6. YM150 Dose Z, once daily (Experimental)
  Interventions: Drug: YM150
- 7. Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: YM150 — oral
  Arms: 1. YM150 Dose V, twice daily; 2. YM150 Dose W, once daily; 3. YM150 Dose X, twice daily; 4. YM150 Dose Y, once daily; 5. YM150 Dose Y, twice daily; 6. YM150 Dose Z, once daily
Drug: Placebo — oral
  Arms: 7. Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of various doses of YM150 (the experimental drug) in the prevention of ischemic vascular events in subjects with recent acute coronary syndromes.

ELIGIBILITY:
Inclusion Criteria:

* has a diagnosis of STE-ACS, NSTE-ACS as index event according to accepted guidelines such as the ESC or AHA guidelines
* has elevated cardiac biomarkers

Exclusion Criteria:

* is planned for myocardial revascularization (e.g., Coronary Artery Bypass Graft (CABG) or elective or staged PCI) or any other invasive procedure with increased risk for bleeding (i.e. elective surgical procedures) within 60 days after randomization
* has had recent stroke or TIA ≤ 12 months prior to index event
* has persistent BP of 160 mmHg systolic or higher and/or 100 mmHg diastolic or higher at baseline with or without medication
* has participated in another clinical trial of an investigational drug (including placebo) or device within 30 days (or the limit set by national law, whichever is longer) of signing informed consent for the present study
* has participated in any YM150 clinical trials
* requires ongoing parenteral or oral anticoagulant therapy
* has active bleeding or is in the opinion of the investigator at high risk of bleeding during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1276 (Actual)
Dates: Start 2009-09; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Incidence of Major and Clinically Relevant Non Major bleeding events according to International Society of Thrombosis and Hemostasis (ISTH) definition | 6 Months

SECONDARY OUTCOMES:
Incidence of Major and Clinically Relevant Non Major bleeding events | 30 Days

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Europe B.V.
Locations (113):
- Argentina (3):
  - Buenos Aires
  - Corrientes
  - Salta
- Australia (2):
  - Concord
  - Douglas
- Belgium (6):
  - Aalst
  - Bonheiden
  - Brussels
  - Genk
  - Leper
  - Ottignies
- Brazil (7):
  - Brasília
  - Porto Alegre
  - Recife
  - Salvador
  - São José
  - São Paulo
  - Uberlândia
- Canada (6):
  - Cambridge
  - Hamilton
  - Laval
  - Longueuil
  - Montreal
  - Saint-Jérôme
- Colombia (4):
  - Barranquilla
  - Bogotá
  - Cartagena
  - Floridablanca
- Czechia (10):
  - Beroun
  - Brno
  - Jihlava
  - Kladno
  - Liberec
  - Pardubice
  - Prague
  - Sternberk
  - Vsetín
  - Zlín
- Copenhagen, Denmark
- Paris, France
- Germany (5):
  - Bad Nauheim
  - Dresden
  - Freiburg im Breisgau
  - Kassel
  - Neuss
- Hungary (8):
  - Balatonfüred
  - Budapest
  - Debrecen
  - Miskolc
  - Nyíregyháza
  - Szeged
  - Székesfehérvár
  - Zalaegerszeg
- India (7):
  - Ahmedabad
  - Hyderabaad
  - Mangalore
  - Nagpur
  - New Delhi
  - Tamil Nadu
  - Tirupati
- Mexico (5):
  - Burócratas del Estado
  - Guadalajara
  - Mérida
  - Morelia
  - Zapopan
- Netherlands (7):
  - 's-Hertogenbosch
  - Amsterdam
  - Heerlen
  - Helmond
  - Leeuwarden
  - Nijmegen
  - Oss
- Poland (6):
  - Bialystok
  - Elblag
  - Gdansk
  - Inowrocław
  - Krakow
  - Przemyśl
- Romania (7):
  - Baia Mare
  - Brăila
  - Bucharest
  - Craiova
  - Oradea
  - Târgovişte
  - Târgu Mureş
- Russia (7):
  - Chelyabinsk
  - Kemerovo
  - Moscow
  - Saratov
  - Tomsk
  - Tyumen
  - Yaroslavl
- Slovakia (4):
  - Martin
  - Nitra
  - Rimavská Sobota
  - Ružomberok
- South Africa (9):
  - George
  - Johannesburg
  - Kuilsriver
  - Parow
  - Pinelands
  - Tongaat
  - Umhlanga
  - Western Cape
  - Worcester
- South Korea (5):
  - Busan
  - Gwangju
  - Gyeonggi-do
  - Inchon
  - Seoul
- Ukraine (3):
  - Kharkiv
  - Kyiv
  - Zaporizhzhya

REFERENCES:
- [Derived] Steg PG, Mehta SR, Jukema JW, Lip GY, Gibson CM, Kovar F, Kala P, Garcia-Hernandez A, Renfurm RW, Granger CB; RUBY-1 Investigators. RUBY-1: a randomized, double-blind, placebo-controlled trial of the safety and tolerability of the novel oral factor Xa inhibitor darexaban (YM150) following acute coronary syndrome. Eur Heart J. 2011 Oct;32(20):2541-54. doi: 10.1093/eurheartj/ehr334. Epub 2011 Aug 30. PMID 21878434